CLINICAL TRIAL: NCT05370716
Title: A Randomized, Open-label, Multiple-dose, Parallel Study to Compare the Pharmacokinetics and to Evaluate Drug-Drug Interaction of "CG-651" in Healthy Volunteers
Brief Title: Drug-Drug Interaction Study of "CG-651" in Healthy Volunteer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: CrystalGenomics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CG100651-1-01
Record Dates: First submitted 2019-12-03; First posted 2022-05-11 (Actual); Last update posted 2022-05-31 (Actual); Status verified 2022-05

CONDITIONS: Healthy
MeSH Terms: interventions — CG100649; Pregabalin

STUDY DESIGN:
Intervention Model Description: * Group A: Pregabalin + Polmacoxib
  * Group B: Polmacoxib
  * Group C: Pregabalin
Masking Description: None (open label)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A (Experimental): Pregabalin + Polmacoxib
  Interventions: Drug: Polmacoxib; Drug: Pregabalin
- Group B (Active Comparator): Polmacoxib
  Interventions: Drug: Polmacoxib
- Group C (Active Comparator): Pregabalin
  Interventions: Drug: Pregabalin

INTERVENTIONS:
Drug: Polmacoxib — Polmacoxib
  Arms: Group A; Group B
Drug: Pregabalin — Pregabalin
  Arms: Group A; Group C

SUMMARY:
This is randomized , open-label, multiple-dose, parallel study to compare the pharmacokinetics and to evaluate Drug-Drug Interaction of "CG-651" in healthy volunteers.

DETAILED DESCRIPTION:
Total of 39 health volunteers will be randomized to receive either of Group A,B or C. (13 subjects each)

[Group A] Pregabalin+ Polmacoxib. [Group B] Polmacoxib [Group C] Pregabalin

ELIGIBILITY:
Key Inclusion Criteria:

* Adequate Biochemistry, Urinalysis, Serology and so on.
* Subject who understand the objective, method of the study and the characteristics of investigational drug and expected adverse events and provide written informed consent prior to study participation.
* Negative pregnancy test (hCG) and agree to contraception during the trial.

Key Exclusion Criteria:

* History of hypersensitivity to investigational products.
* History of hypersensitivity or allergic reaction to sulfonamide.
* Patients with a history of asthma, acute rhinitis, non specific polyps, angioedema, urticaria or allergic reactions to aspirin or other nonsteroidal anti-inflammatory analgesics(including COX-2 inhibitors)
* Any other reason or situations that the investigator decides the patient is not eligible to participate the clinical trial.

Ages: 19 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 47 (Actual)
Dates: Start 2019-11-11 (Actual); Primary Completion 2020-04-30 (Actual); Study Completion 2020-05-19 (Actual)

PRIMARY OUTCOMES:
Cmax of polmacoxib and pregabalin | upto 4 weeks
  Maximum Observed Plasma Concentration
AUC of polmacoxib and pregabalin | upto 4 weeks
  Area Under the Concentration-Time Curve
The Number of Participants Who Experienced Adverse events (AEs) | upto 4 weeks
  A non-serious adverse event is any untoward medical occurrence. A serious adverse event is any adverse event that meets one or more of the following: results in death; is life-threatening; requires inpatient hospitalization or prolongation of existing hospitalization; results in persistent or significant disability/incapacity; is a congenital anomaly/birth defect; requires intervention to prevent permanent impairment or damage.

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, South Korea